CLINICAL TRIAL: NCT00929448
Title: The Predictive Value of Clinical and Immunological Factors in the Development of Pneumonia After Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Royal Alexandra Hospital (Other)
Responsible Party: Principal Investigator, Demetrios J. Kutsogiannis, MD, MHS, FRCPC, Royal Alexandra Hospital
Other Study IDs: iTBI2009
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Immunoglobulin

SUMMARY:
The development of pneumonia and other infections is one of the most common complications of a traumatic brain injury (TBI). Prior studies have also found that patients suffering from TBI also develop immune dysfunction consistent with an immunosuppressed state shortly after the traumatic event. Specifically, it has been shown that patients with a TBI have impaired delayed type hypersensitivity (DTH), cellular immunity and humoral immunity. The humoral arm of the immune system is particularly involved in defending the host against extracellular bacteria and is primarily composed of B-cells, immunoglobulins and complement. Surgery and trauma impair the clonal expansion of antibody producing B lymphocytes causing hypogammaglobulinemia, through a mechanism involving T lymphocytes. In addition, during the systemic inflammatory process, pro-inflammatory cytokines such as tumor necrosis factor alpha (TNF-alpha), interleukin 1 (IL-1beta) and interleukin 6 (IL-6) are released. Nuclear factor kappa beta (NF-kB) is a transcriptional regulatory protein that is involved in the expression of proinflammatory cytokines and appears to act at a critical step in the transcription of many proinflammatory genes.

The hypothesis of this study is that the hypogammaglobulinemia from the immune dysfunction and the induction of NF-kB from the inflammatory process are, in part, responsible for the development of pneumonia and other infectious complications identified after TBI. This study has two specific aims: The primary specific aim of this study is to determine the association between serum immunoglobulin or NF-kB levels and the development of pneumonia in patients suffering from traumatic brain injury (TBI). The secondary specific aim of this study is to determine the relative contribution of clinical variables such as APACHE II-III Score and Injury Severity Score as compared to immunological variables (serum immunoglobulins and NF-kB) to the development of pneumonia in patients suffering from TBI.

ELIGIBILITY:
Inclusion Criteria:

* > 18 yrs
* Admitted to ICU in Capital Health region with a TBI and > 1 of the following:
* An initial resuscitated (Sys BP>90 mmHg and O2 Sat >90%) GSC of ≤ 8
* A post resuscitation (Sys BP>90 mmHg and O2 Sat >90%) GCS at presentation to the hospital of ≤ 8 in the absence of sedation
* A post resuscitation (Sys BP>90 mmHg and O2 Sat >90%) GCS within 72 hrs of hospital admission of ≤ 8 in the absence of sedation
* Intracranial pressure monitoring
* Decompressive craniectomy
* Presence of subfalcine, uncal, or supratentorial herniation either clinically or radiologically

Exclusion Criteria:

* Longer than 5 days since ictus of TBI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2008-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study will be the development of the composite of either early onset pneumonia (EOP) or ventilator associated pneumonia (VAP | baseline, d4, d7, d10, d14

SECONDARY OUTCOMES:
Secondary outcomes will include ICU and hospital mortality and LOS, duration of mechanical ventilation, Glasgow Outcome Score (GOS) at hospital discharge and at 6-months, and 1-year. | hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Demetrios Kutsogiannis, MD, Principal Investigator — Royal Alexandra Hospital
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada